CLINICAL TRIAL: NCT01842581
Title: A Multicenter, Randomized, Open-Label, Active-Controlled, Trial to Evaluate the Safety and Efficacy of Rifaximin 550 mg With and Without Lactulose in Subjects With a History of Recurrent Overt Hepatic Encephalopathy
Brief Title: The Safety/Efficacy of Rifaximin With/Without Lactulose in Participants With A History of Recurrent Hepatic Encephalopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFHE4044
Record Dates: First submitted 2013-04-16; First posted 2013-04-29 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Hepatic Encephalopathy; Cirrhosis
Keywords: Liver Failure; Hepatic Insufficiency; Liver Diseases; Brain Diseases; Rifaximin; Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis; Liver Failure; Hepatic Insufficiency; Liver Diseases; Brain Diseases | interventions — Rifaximin; Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rifaximin 550 mg BID (Experimental): Participants will receive rifaximin 550 milligrams (mg) tablet orally twice daily (BID) for 24 weeks.
  Interventions: Drug: Rifaximin
- Rifaximin 550 mg BID + Lactulose (Experimental): Participants will receive rifaximin 550 mg tablet orally BID with lactulose solution for 24 weeks. Lactulose dose will be self-titrated by the participant to produce 2 to 3 soft stools per day.
  Interventions: Drug: Rifaximin; Drug: Lactulose

INTERVENTIONS:
Drug: Rifaximin — Rifaximin will be administered per the dose and schedule specified in the arms.
  Other Names: Xifaxan®
Drug: Lactulose — Laculose will be administered per the schedule specified in the respective arm.
  Arms: Rifaximin 550 mg BID + Lactulose

SUMMARY:
The purpose of the study is to evaluate if rifaximin alone or rifaximin plus lactulose delays the onset of hepatic encephalopathy (HE) in participants with cirrhosis who have had a previous episode of HE.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females greater than or equal to (≥) 18 years old.
* In remission from demonstrated overt HE (Conn score 0 or 1).
* Have had one or more episodes of overt HE associated with cirrhosis within 6 months prior to screening visit (Day -7 to -1).
* Participant has a close family member or other personal contact who is familiar with the participant's HE and can provide continuing oversight to the participant and is willing to perform as caregiver for the participant during the conduct of the trial.

Exclusion Criteria:

* Participant has been diagnosed with human immunodeficiency virus (HIV) as determined by medical history.
* History of tuberculosis infection.
* Participant has been diagnosed with chronic respiratory insufficiency.
* Participant has been diagnosed with a current infection for which they are currently taking oral or parenteral antibiotics.
* Renal insufficiency requiring routine dialysis.
* Participant has an active spontaneous bacterial peritonitis(SBP) infection.
* Intestinal obstruction or inflammatory bowel disease.
* Participant has active malignancy within the last 5 years prior to screening visit, except basal cell carcinoma of the skin, or if female, in situ cervical carcinoma that has been surgically excised.
* Current gastrointestinal (GI) bleeding or has a history of a GI hemorrhage of sufficient severity to require hospitalization and a transfusion of ≥2 units of blood within 3 months prior to screening visit.
* Participant is anemic, as defined by a hemoglobin of less than (<) 8 grams/deciliter (g/dL).
* Scheduled to receive a liver transplant within 1 month of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2014-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (43):
- United States (43):
  - Banner Research, Phoenix, Arizona
  - Southern California Liver Centers, Coronado, California
  - UCSF/Fresno - CRMC, Fresno, California
  - UCSD Clinical & Translational Research Institute, La Jolla, California
  - Salix Site, Long Beach, California
  - Inland Empire Liver Foundation, Rialto, California
  - Salix Site, Riverside, California
  - Salix Site, San Diego, California
  - Salix Site, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - South Denver GI, Englewood, Colorado
  - University of Florida Hepatology, Gainesville, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Gastroenterology Associates, Macon, Georgia
  - Salix Site, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Central Iowa Hospital Corp, Des Moines, Iowa
  - Salix Site, Jefferson, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - The Center for Liver and Biliary Disease, Baltimore, Maryland
  - Brigham and Women's Hospital Division of Gastroenterology & Hepatology, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Research Institute, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Univ. of Nebraska Medical Center, Omaha, Nebraska
  - Concorde Medical Group PLLC, New York, New York
  - New York University Medical Center, New York, New York
  - Salix Site, New York, New York
  - Columbia University Medical Ctr. Center for Liver Disease & Transplantation, New York, New York
  - University of Rochester Strong Memorial Hospital, Rochester, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - UNC School of Medicine/Division of Gastroenterology and Hepatology, Chapel Hill, North Carolina
  - Carolina Medical Center, Charlotte, North Carolina
  - Integris Nazh Zuhdi Transplant Institute, Oklahoma City, Oklahoma
  - Albert Einstien Medical Center, Philadelphia, Pennsylvania
  - Research Specialists of Texas, Houston, Texas
  - Amcare Research Inc, Houston, Texas
  - Salix Site, Odessa, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Methodist Hospital, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - VCU/MCV Health Systems, Richmond, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 222 participants with cirrhosis and in remission from demonstrated hepatic encephalopathy (HE) were enrolled and randomized in a 1:1 ratio to either Rifaximin 550 mg BID or Rifaximin 550 mg BID + Lactulose treatment arm.
Groups:
- Rifaximin 550 mg BID: Participants received rifaximin 550 milligrams (mg) tablet orally twice daily (BID) for 24 weeks.
- Rifaximin 550 mg BID + Lactulose: Participants received rifaximin 550 mg tablet orally BID with lactulose solution for 24 weeks. Lactulose dose was self-titrated to produce 2 to 3 soft stools per day.
Period: Overall Study
Arm/Group | Rifaximin 550 mg BID | Rifaximin 550 mg BID + Lactulose
Started | 113 | 109
Received at Least 1 Dose of Study Drug | 113 | 108
Completed | 69 | 79
Not Completed | 44 | 30
Not completed — Adverse Event | 6 | 4
Not completed — HE breakthrough | 26 | 13
Not completed — Liver transplant | 2 | 0
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Other than specified | 3 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Rifaximin 550 mg BID: Participants received rifaximin 550 mg tablet orally BID for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Rifaximin 550 mg BID | Rifaximin 550 mg BID + Lactulose | Total
Number analyzed (Participants) | 113 | 108 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.51) | 58.8 (9.49) | 58.4 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 38 | 82
  Male | 69 | 70 | 139
Lactulose Usage Prior to First Dose [Count of Participants; unit: Participants]
  Yes | 100 | 100 | 200
  No | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting a First Breakthrough HE Episode
Description: A breakthrough HE episode was defined as an increase of the Conn score to Grade greater than or equal to (≥) 2 (ie, 0 or 1 to ≥ 2). Conn score is widely used as a measure of mental state in HE. The scale used in Conn scoring system include: Grade 0=No personality or behavioral abnormality; Grade 1=Trivial lack of awareness, euphoria, or anxiety; shortened attention span, impairment of addition or subtraction; Grade 2=Lethargy, disorientation for time, obvious personality change, inappropriate behaviour; Grade 3=Somnolence to semi-stupor, responsive to stimuli, confused, gross disorientation, bizarre behaviour; Grade 4=Coma, unable to test mental state. The time to the first breakthrough HE episode was defined as the duration between the date of first dose of study drug and the date of first breakthrough HE episode. Number of participants reporting a first breakthrough HE episode during randomization to Month 6 is presented.
Time Frame: From randomization (Day 1) up to Day 170
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin 550 mg BID | Rifaximin 550 mg BID + Lactulose
Number analyzed (Participants) | 113 | 108
Participants | 28 | 15
Statistical Analysis 1: Comparison: Rifaximin 550 mg BID vs Rifaximin 550 mg BID + Lactulose; Hazard ratio estimate (hazard of breakthrough HE for rifaximin compared to rifaximin + lactulose) obtained from Cox proportional hazards model with effect for treatment, stratified by analysis region; Test type: Non-Inferiority — Threshold for significance=upper bound of the 2-sided 95% confidence interval (CI) for hazard ratio less than (<) 1.56; p = 0.0359, Score statistics; Hazard Ratio (HR) = 1.959, 95% CI 2-sided [1.045 to 3.672]

2. Secondary Outcome: Number of Participants Who Were Hospitalized Due to HE Episode
Description: An HE-related hospitalization was defined as a hospitalization directly resulting from HE, or when HE events occurred during hospitalization. The time to first HE-related hospitalization was defined as the duration between the date of first dose of study drug and the date of first HE-related hospitalization. Number of participants who were hospitalized due to HE episode during randomization to Month 6 is presented.
Time Frame: From randomization (Day 1) up to Day 170
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin 550 mg BID | Rifaximin 550 mg BID + Lactulose
Number analyzed (Participants) | 113 | 108
Participants | 23 | 14
Statistical Analysis 1: Comparison: Rifaximin 550 mg BID vs Rifaximin 550 mg BID + Lactulose; Analysis was performed using log-rank test stratified by analysis region. Hazard ratio estimate (hazard of breakthrough HE for rifaximin compared to rifaximin + lactulose) obtained from Cox proportional hazards model with effect for treatment, stratified by analysis region; Test type: Superiority — 2-sided test at a significance level of 0.05; p = 0.0985, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 1.739, 95% CI 2-sided [0.894 to 3.382]

3. Secondary Outcome: Number of Participants Who Died Due to Any Reason
Time Frame: From randomization (Day 1) up to end of study (Day 186)
Population: Safety population was the same as the ITT population that included randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin 550 mg BID | Rifaximin 550 mg BID + Lactulose
Number analyzed (Participants) | 113 | 108
Participants | 2 | 2

4. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAE was defined as an AE that occurred from first dose of study drug until last dose of study drug plus 5 days (for non-fatal AEs) or plus 30 days (for fatal AEs).A summary of non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: From randomization (Day 1) up to end of study (Day 186)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin 550 mg BID | Rifaximin 550 mg BID + Lactulose
Number analyzed (Participants) | 113 | 108
Participants | 99 | 81

5. Other Pre Specified Outcome: Change From Baseline in Total Chronic Liver Disease Questionnaire (CLDQ) Score at Day 170
Description: CLDQ was used to measure health-related quality of life. CLDQ includes 29 items in the following 6 domains: abdominal symptoms (3 items), fatigue (5 items), systemic symptoms (5 items), activity (3 items), emotional function (8 items), and worry (5 items). All items were measured on a 7-point Likert scale, ranging from 0 to 6 with higher values indicating better quality of life. Each domain score of CLDQ was calculated as the mean of the responses of items in that domain. Overall CLDQ score was obtained by adding scores for each item and dividing by the total number of items. Overall CLDQ score ranged from 0 (most impairment) to 6 (least impairment) with higher scores indicating better quality of life. If at least half of the items were non-missing for a domain, mean values of the non-missing items for that domain were used as imputed values for missing values. If more than half of the items in a domain were missing, no values were imputed and domain score was considered as missing.
Time Frame: Baseline, Day 170
Population: ITT population included all randomized participants who received at least 1 dose of study drug. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rifaximin 550 mg BID | Rifaximin 550 mg BID + Lactulose
Number analyzed (Participants) | 113 | 108
units on a scale
  Baseline | 4.13 (1.110) | 4.26 (1.197)
  Change at Day 170: number analyzed (Participants) | 112 | 100
  Change at Day 170 | 0.29 (0.860) | 0.08 (1.055)

6. Other Pre Specified Outcome: Change From Baseline in Critical Flicker Frequency (CFF) at Day 170
Description: The critical flicker frequency (CFF), a validated assessment of neurological function was assessed using a specialized CFF instrument. The CFF is the frequency at which the participant observes a constant light transition to a flickering light and was measured in Hertz. The CFF was measured on a continuous scale and was the mean of 8 separate fusion-to-flicker transition tests performed in rapid succession. Increases in CFF results represent improvement in neurological function in participants with HE.
Time Frame: Baseline, Day 170
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hertz
Arm/Group | Rifaximin 550 mg BID | Rifaximin 550 mg BID + Lactulose
Number analyzed (Participants) | 113 | 108
hertz
  Baseline | 35.14 (7.767) | 34.64 (7.290)
  Change at Day 170: number analyzed (Participants) | 111 | 101
  Change at Day 170 | 1.09 (7.266) | 2.10 (6.699)

ADVERSE EVENTS:
Time Frame: From randomization (Day 1) up to end of study (Day 186)
Description: Safety population was the same as the ITT population that included randomized participants who received at least 1 dose of study drug.
Arm/Group | Rifaximin 550 mg BID | Rifaximin 550 mg BID + Lactulose
Serious Adverse Events (participants affected / at risk) | 43/113 | 35/108
Other Adverse Events (participants affected / at risk) | 68/113 | 53/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin 550 mg BID (N=113) | Rifaximin 550 mg BID + Lactulose (N=108)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 3 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 2 | 2
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 4
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Alcoholic seizure (Nervous system disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 21 | 10
Presyncope (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 6 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Liver transplant (Surgical and medical procedures) | 2 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin 550 mg BID (N=113) | Rifaximin 550 mg BID + Lactulose (N=108)
Anaemia (Blood and lymphatic system disorders) | 6 | 2
Abdominal distension (Gastrointestinal disorders) | 3 | 7
Abdominal pain (Gastrointestinal disorders) | 8 | 8
Ascites (Gastrointestinal disorders) | 7 | 10
Constipation (Gastrointestinal disorders) | 18 | 9
Diarrhoea (Gastrointestinal disorders) | 5 | 13
Flatulence (Gastrointestinal disorders) | 1 | 6
Nausea (Gastrointestinal disorders) | 16 | 11
Vomiting (Gastrointestinal disorders) | 6 | 6
Asthenia (General disorders) | 6 | 2
Fatigue (General disorders) | 16 | 9
Oedema peripheral (General disorders) | 19 | 15
Jaundice (Hepatobiliary disorders) | 4 | 6
Urinary tract infection (Infections and infestations) | 12 | 5
Decreased appetite (Metabolism and nutrition disorders) | 8 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 11
Headache (Nervous system disorders) | 7 | 5
Anxiety (Psychiatric disorders) | 6 | 10
Depression (Psychiatric disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 13 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Pruritus generalised (Skin and subcutaneous tissue disorders) | 11 | 6

LIMITATIONS AND CAVEATS:
The rifaximin monotherapy arm included a subset of rifaximin/lactulose dependent participants for whom lactulose was withdrawn upon randomization (88.5% of participants in that group), which led to earlier HE breakthrough in this subset.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.